CLINICAL TRIAL: NCT05669716
Title: Adolescent Vaping Characterization and Parent Views on Adolescent Vaping Protocol
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator is leaving NIDA.
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001196; 001196-DA
Record Dates: First submitted 2022-12-30; First posted 2023-01-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Vaping Teens
Keywords: Vape; Nicotine; Teen; Drug Use; Natural History
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- parents of teens who vape: 400 parent participants, defined as an adult who identifies as parenting an adolescent aged 13-17 whom they know/suspect is vaping.
- teens who formerly vaped: Adolescents N=400 (formerly vaped)
- teens who never vaped: Adolescents N=400 (never vaped).
- teens who vape: adolescent participants (minor subjects), comprised of N=400 (currently vaping, defined as vaping at least one day in the previous 30-day period

SUMMARY:
Background:

The use of electronic cigarettes (vaping) has increased among adolescents over the past decade. Vaping raises many health concerns. People who vape inhale toxic chemicals. Vaping is also linked with mental health issues, such as depression and suicide risk. In one survey, 85% of young adults reported that they used both vaping and tobacco products; the primary reason they cited for using these products was stress.

Objective:

This natural history study will survey adolescents and their parents about their attitudes toward vaping.

Eligibility:

People aged 13 to 18, including those who vape; those who once vaped; and those who have never vaped. Parents of people aged 13 to 18 who are known or suspected of vaping are also needed.

Design:

Participants will take a survey. They will use their own smartphone, computer, or tablet to answer questions. The survey will take about 20 minutes. Their answers will be anonymous.

Teenage participants will answer questions on different topics:

Vaping habits, such as when and how they vape.

Drug use, including nicotine, cannabis, and alcohol.

Mood issues, such as depression, anxiety, and stress.

Social influences on vaping, including perceived attitudes of parents and peers.

Other leisure habits, including online gaming and use of social media.

Parents will answer similar questions.

A phone number and links will be given to participants who need help for suicidal thoughts. Other links will be given to those who want help with parenting resources or aids to quit vaping.

Participants may be invited to take part in an 8-week course on mindfulness-based stress reduction.

Participants who finish the survey will receive 10 dollars.

...

DETAILED DESCRIPTION:
Study Description: This protocol will explore characteristics of adolescents who vape and the attitudes of adolescents and parents of adolescents who vape towards adolescent vaping, focusing on the Baltimore area. Hypotheses: (Adolescent) Currently vaping adolescents will not view vaping as a problem for which they seek help and will have more mental health symptoms than non-vaping adolescents, while non-vaping adolescents will view vaping more negatively with formerly vaping adolescents scoring between the currently vaping and non-vaping adolescent groups. (Parent) Parents who vape will be more likely to approve of their adolescent s vaping than non-vaping parents.

Objectives:

Primary Objective: To characterize adolescent vaping patterns, overall drug use, perceived stress, and awareness of mindfulness meditation.

Secondary Objectives: To characterize the mental health symptoms of currently vaping, formerly vaping and non-vaping adolescents, and to characterize parent attitudes towards their adolescent s vaping.

Endpoints:

Primary Endpoint: An adequate description of adolescent vapers habits and attitudes towards their vaping.

Secondary Endpoints: An adequate comparison of adolescent vapers, former vapers and non-vapers and of parental attitudes towards adolescent vapers.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must:

Be an adolescent age 13-18 and in grades 8-12 or the summer after graduation, OR an adult who identifies as parenting an adolescent aged 13-18 and in grades 8-12 or the summer after graduation whom they know/suspect is vaping or never has vaped. All participants must be willing to complete the survey to the end.

EXCLUSION CRITERIA:

Non-English speakers cannot participate in this study. Justification: The questionnaires from which the survey is constructed are not all validated in languages other than English. We do not have the resources to translate the consent and surveys.

Those who cannot demonstrate understanding of the purpose of the survey by answering questions after a brief explanation will be excluded. Justification: The ability to understand the purpose of the survey is required in order to provide informed consent to participate and to be able to provide meaningful answers to the survey questions.

Ages: 13 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and parent participants will be enrolled in the survey through the internet, via their own smartphone/computer/tablet device.
Sampling Method: Non-Probability Sample
Enrollment: 726 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Attitude toward vaping | at time of survey
  An adequate description of adolescent vapers habits and attitudes towards their vaping.

SECONDARY OUTCOMES:
characteristics of parents of teens who vape | at time of survey
  parental attitudes towards adolescent vapers.
comparison of vaping and non-vaping teens on mental health and other drug use | at time of survey
  An adequate comparison of adolescent vapers, former vapers and non-vapers on mental health and other drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Jo Salmeron, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We plan to share data as specified in the protocol and potentially through future data transfer agreement(s). Any shared data will be stripped of identifiers prior to release for sharing. Deidentified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place. Outside of the data sharing plan already specified in the protocol (in what would be outline in a future data sharing agreement), we have not yet finalized decisions on types of supporting information that will be shared, IPD Sharing Time Frame, IPD Sharing Access Criteria for other future data sharing agreements.